CLINICAL TRIAL: NCT05069194
Title: Study on the Etiology, Risk Factors and Pathogenesis ofCOPD Based on Clinical Bioinformatics
Brief Title: Study on the Etiology, Risk Factors and Pathogenesis of COPD Based on Clinical Bioinformatics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); The Second Affiliated Hospital of Fujian Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Xibei Hospital (Other); Henan Provincial People's Hospital (Other); Shenzhen University (Other); Shantou University Medical College (Other); Shanghai Minhang Central Hospital (Other); Shanghai Fengxian District Central Hospital (Other); Sun Med IT(ShangHai) Co. Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2016YFC1304000
Record Dates: First submitted 2019-07-15; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood，bronchial epithelium,sputum,bronchial alveolar lavage,lung tissue ,mouse
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD: Patients with chronic obstructive pulmonary disease
- High Risk: People who do not suffer from COPD, but have high risk factor for COPD.
- Health: People who do not suffer from COPD and do not have a high risk factor for COPD either.

SUMMARY:
The risk factors and causes of chronic obstructive pulmonary disease（COPD）are not clear, so the prevalence of COPD is high and the prevention effect is not good. Because the pathogenesis of COPD is not completely elucidated, the diagnosis and classification of COPD are inaccurate which resulting in poor efficacy of treatment. Therefore, it is of great scientific and clinical significance to find out the risk factors and causes of COPD, to clarify its pathogenesis, to put forward the prevention and early intervention measures of COPD, to warn the occurrence of COPD, to predict the deterioration of the disease, to reduce the occurrence of COPD and to slow down the progress of COPD.

The project establishes a cohort of COPD people，high-risk group and the healthy group. The project studys the risk factors, etiology and pathogenesis of COPD. The project studys the interaction between genetic factors and environmental factors on COPD and its effect on pathogenesis, progression and outcome of COPD.

DETAILED DESCRIPTION:
The project establishes the data base and specimen bank for COPD.Then clinical bioinformatics technology is uesd to analyze the clinical information and epidemiological information. In the same time, Omics methods are used to study COPD-related genes and biomarkers . Finally, a multi-factor risk factor model for the occurrence and development of COPD is established by combining clinical information, epidemiological information and biomics results.

ELIGIBILITY:
Inclusion Criteria:

① Inclusion criteria for patients with COPD:

* Over 18 years of age.
* FEV1 / FVC< 70% was the diagnostic criterion for COPD after inhaling bronchodilators.

  ② Inclusion criteria for high-risk subjects:
* Over 18 years of age.
* Physical examination and routine laboratory tests were normal.
* Chest CT to exclude other pulmonary diseases.
* Lung function does not meet the diagnostic criteria for COPD.
* having one of the following risk factors: A. Smoking: current smokers, smoking index (number of years of smoking × number of cigarettes per day)≥ L.

B. Biofuel exposure: Subjects frequently use charcoal, wood, and animal dung for home heating and cooking Or crops are defined as having a history of exposure to biofuels. C. Dust and chemical exposure: mining, quarrying, casting, grain dust, paint, chemicals and others (including non-return) In the above categories of self-reported) occupational dust or gas smoke exposure for more than 1 year.

③ Inclusion criteria of healthy control subjects:

* Over 18 years of age.
* Physical examination and routine laboratory tests were normal.
* Chest CT to exclude other pulmonary diseases.
* Lung function does not meet the diagnostic criteria for COPD.
* No risk factors (including smoking, biofuel exposure, dust or chemical exposure).

Exclusion Criteria:

* History of other chronic lung diseases, such as bronchiectasis, pulmonary interstitial fibrosis, etc.
* History of acute lung disease within 3 months.
* History of malignant tumor.
* Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from Shanghai City, Wenzhou City, Quanzhou City, Zhengzhou City and Xi'an City.
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2017-12-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk factors and pathogenesis of of COPD | From date of participation in project until December 31, 2022
  1. To establish a cohort of copd patients and high-risk population;
  2. To establish a multi-factor risk factor model for copd, and screen 5-10 risk factors related to the occurrence and development of COPD.

SECONDARY OUTCOMES:
Clinical bioinformatics database for COPD | From date of participation in project until December 31, 2022
  1. To find 1-2 susceptibility genes closely related to COPD through gene and epigenetic studies combined with clinical bioinformatics analysis and genomic research ;
  2. To find 3-5 biomarkers closely related to COPD through protein and metabolomics studies as well as clinical bioinformatics analysis.
Biological library of COPD | From date of participation in project until December 31, 2022
  1. To verify the identified susceptibility genes and biomarkers in the existing COPD cohort, and then expand to be verified outside the cohort, to verify 5-7 related susceptibility genes and biomarkers;
  2. To further explore the pathogenesis of COPD by conducting preliminary mechanism studies on the discovered susceptibility genes and biomarkers combined with big data analysis;
  3. To build a unified copd data collection and sharing platform between local hospitals to achieve real-time monitoring of statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: ChengShui Chen, Study Chair — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The first affiliated hospital of wenzhou medical university, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided